CLINICAL TRIAL: NCT01101867
Title: Prandial Insulin Dosing Using the Carbohydrate Counting Technique in Hospitalized Patients With Diabetes
Brief Title: Prandial Insulin Dosing in Hospitalized Patients
Acronym: ICHO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kathleen Dungan (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Kathleen Dungan, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Novo Nordisk xxxx
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Diabetes; Admitting Hospital; Non-critically Ill
Keywords: diabetes; glucose; hospital
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspart flexible dose (Experimental): aspart dose determined based upon carbohydrate intake.
  Interventions: Drug: Aspart flexible dose
- Aspart fixed dose (Active Comparator): fixed meal dose of aspart (based upon weight or total daily insulin dose)
  Interventions: Drug: Aspart fixed dose

INTERVENTIONS:
Drug: Aspart fixed dose — fixed dose
  Other Names: Novolog
  Arms: Aspart fixed dose
Drug: Aspart flexible dose — dose based upon carbohydrate intake and total daily requirements
  Other Names: Novolog
  Arms: Aspart flexible dose

SUMMARY:
The purpose of this study is to determine whether mealtime insulin results in better control of blood sugar than a fixed meal dose in hospitalized patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether mealtime insulin, dosed to match the intake of carbohydrates (starches or sugars) results in better control of blood sugar than a fixed meal dose in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* general medical or minor surgical hospitalized patients
* type 2 diabetes
* blood glucose 150-400 on at least 2 occasions within 24 hours or requiring at least 20 units of insulin/day in the 24 hours prior to enrollment

Exclusion Criteria:

* • Major surgery, occurring within the previous 2 weeks or planned within 72 hours of study entry, including cardiothoracic, neurosurgical, and open intra-abdominal procedures (in particular, any surgery lasting over 2 hours).

  * Patients receiving glucocorticoids, total parental nutrition (TPN), or tube feeds.
  * Pregnancy (glucose targets differ in pregnancy). Premenopausal women not on pharmacologic contraceptives, inrauterine device (IUD), or surgical menopause will undergo pregnancy testing.
  * Patients currently on IV insulin (must wait to enroll) or with planned surgical procedures in the next 72 hours for whom intravenous insulin will be likely
  * Prolonged (>24 hour) strict nil per os (NPO-nothing by mouth) status (eg. small bowl obstruction). Liquid or modified consistency diets are acceptable.
  * Patients for whom expected length of stay will be less than 48 hours
  * Patients using subcutaneous insulin pumps
  * Diabetic ketoacidosis
  * End-stage renal disease on dialysis
  * End-stage liver disease with cirrhosis
  * Mental conditions precluding informed consent
  * Potentially sensitive admissions: prisoners, HIV, suicidality
  * Unable to give consent in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Flexible Dose: Insulin Aspart dose is determined based upon carbohydrate intake and is administered immediately post-meal. Prandial insulin was based upon the formula: CIR=400/TDD where CIR refers to the carbohydrate-to-insulin ratio and TDD refers to the total daily calculated dose of insulin (based upon total daily insulin dose or upon weight, depending upon whether a patient is insulin naive or not, respectively).
- Fixed Dose: Fixed meal dose of Insulin Aspart (based upon total daily insulin dose or upon weight, depending upon whether a patient is insulin naive or not, respectively). Half of the TDD was divided into three equal fixed doses given immediately after each meal.
Period: Overall Study
Arm/Group | Flexible Dose | Fixed Dose
Started | 63 | 63
Completed | 62 | 59
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Flexible Dose: aspart dose determined based upon carbohydrate intake.
- Fixed Dose: fixed meal dose of aspart (based upon weight or total daily insulin dose)
- Total: Total of all reporting groups
Arm/Group | Flexible Dose | Fixed Dose | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 49 | 97
  >=65 years | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 56 (12) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 38 | 34 | 72
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126

OUTCOME MEASURES:

1. Primary Outcome: Mean Glucose
Description: Mean glucose was calculated per participant from the average of glucose values over the 7-point (pre- and post-breakfast, lunch, dinner, and bed) glucose profile at day 3
Time Frame: day 3
Population: Data were only available in 79 subjects on day 3 due to hospital discharge or NPO status.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Flexible Dose | Fixed Dose
Number analyzed (Participants) | 42 | 37
mg/dl | 158 (47) | 171 (49)

2. Secondary Outcome: Postprandial Glucose
Description: Mean postprandial glucose was calculated per participant from the average of glucose values (post-breakfast, lunch, dinner) at day 3.
Time Frame: day 3
Population: Data were only available in 79 subjects on day 3 due to hospital discharge or NPO status.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Flexible Dose | Fixed Dose
Number analyzed (Participants) | 42 | 37
mg/dl | 175 (51) | 203 (74)

3. Secondary Outcome: Hypoglycemia
Description: Number of patients with any hypoglycemic event (<70 mg/dl or <40 mg/dl)
Time Frame: 72 hour
Measure: Number; unit: participants
Arm/Group | Flexible Dose | Fixed Dose
Number analyzed (Participants) | 62 | 59
participants | 24 | 14

4. Secondary Outcome: Change in Glucose
Description: Change in mean glucose from day 1 to day 3, measured as difference in mean glucose day 3 minus mean glucose day 1.
Time Frame: 72 hour
Population: intention to treat population
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Aspart Flexible Dose | Aspart Fixed Dose
Number analyzed (Participants) | 42 | 37
mg/dl | -4.2 (35) | -8.1 (54)

5. Secondary Outcome: Treatment Satisfaction
Description: treatment satisfaction questionnaire validated in-hospital, 19 item questionnaire using 0-6 point likert scale, for minimum zero to maximum of 102 points (with 102 indicating best satisfaction). Items are summed to find the total score.
Time Frame: day 3
Population: all participants who completed the survey
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Flexible Dose | Fixed Dose
Number analyzed (Participants) | 50 | 50
points on a scale | 69 (14) | 68 (13)

6. Secondary Outcome: 1,5-anhydroglucitol Change
Description: change in short-term measure of glycemia
Time Frame: day 1 to day 3
Population: subjects with complete data
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Flexible Dose | Fixed Dose
Number analyzed (Participants) | 41 | 32
mcg/ml | 0.41 (2.76) | 0.73 (3.96)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Flexible Dose | Fixed Dose
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 24/62 | 14/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flexible Dose (N=62) | Fixed Dose (N=59)
Hypoglycemia (BG <70 mg/dl) (Endocrine disorders) | 24 | 14

LIMITATIONS AND CAVEATS:
Miscalculation of meal doses, mistimed doses, lack of complete documentation of carbohydrate intake, and dosing conducted by an experienced clinician may have contributed to the findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No